CLINICAL TRIAL: NCT04430127
Title: The Role of Quantitative Measures on Dual-energy CT in the Prediction of Colorectal Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital Fribourgeois (Other)
Responsible Party: Principal Investigator, Malekzadeh, Principal Investigator, Hôpital Fribourgeois
Other Study IDs: 2020-00052
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Adenocarcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal adenocarcinoma: patients with pathology-proved colorectal tumor (detected by optical colonoscopy) who undergo routine thoraco-abdominal DECT for initial staging
  Interventions: Other: No supplementary intervention is performed

INTERVENTIONS:
Other: No supplementary intervention is performed — No supplementary intervention will be applied

SUMMARY:
To demonstrate the potential role of dual-energy computed tomography (DECT) by iodine maps data, aimed at discriminating colon cancer from colon wall pseudo-thickening.

DETAILED DESCRIPTION:
Prospectively, 50 consecutive patients with pathology-proved colorectal tumor (detected by optical colonoscopy) who undergo routine thoraco-abdominal DECT for initial staging in the Department of Radiology at our institution from April 2020, will be included. The exclusion criteria are as follows: patients with body mass index (BMI) above 30 kg/m2, patients with renal insufficiency (estimated glomerular filtration rate < 30 ml/min), allergy to iodinated contrast and a known history of previous abdominal radiotherapy.

All patients will undergo a staging enhanced thoraco-abdominal CT by 256-slices CTs (Revolution CT, GE healthcare) at Fribourg hospital. DECTs will be acquired without an enema, rectal insufflation or oral contrast to have collapsed colorectal wall for further measurements and to simulate routine clinical practice. No additional screening procedures, such as a laboratory or diagnostic tests are necessary for the present study.

Upon acquiring 50 patients, CT quantitative assessments will be performed. Initially, data will be transferred to AW Advantage workstations (GE Healthcare). Thereafter, for each patient, the iodine map images will be created by post-processing by. All CT quantitative measurements will be performed independently by two radiologists. Three regions of interest (ROI) will be applied to colorectal tumor and the normal collapsed colorectal wall (confirmed previously by colonoscopy) and consequently, the mean of these measurements will be reported. These measurements correspond to mean iodine uptake of colorectal tumor and normal collapsed wall, respectively. Finally, the iodine uptake of the tumoral lesion and normal collapsed wall in each patient will be compared to demonstrate the significant difference in iodine uptake. Investigators anticipate that the obtained cut-off value will be a new benchmark in clinical practice, to exclude the colorectal tumors on non-prepared collapsed colon wall and eliminate the need for a complementary colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

. pathology-proved colorectal tumor

Exclusion Criteria:

* BMI above 30 kg/m2
* renal insufficiency (estimated glomerular filtration rate < 30 ml/min),
* allergy to iodinated contrast, and a
* known history of previous abdominal radiotherapy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathology-proved colorectal tumor (detected by optical colonoscopy) who undergo routine thoraco-abdominal DECT for initial staging in the Department of Radiology at our institution from April 2020
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference of iodine uptake | 3.11.2021
  Difference of iodine uptake between colorectal tumor and pseudo-thickened colorectal wall on DECT

CONTACTS AND LOCATIONS:
Locations (1):
- Sonaz Malekzadeh, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No